CLINICAL TRIAL: NCT00387621
Title: To Define in Normal Controls, Human Preclinical Systolic Dysfunction (PSD) and Preclinical Diastolic Dysfunction (PDD) the Actions of Acute Subcutaneous Nesiritide (BNP) on the Cardiorenal and Humoral Function and the Integrated Response to Acute Sodium Loading
Brief Title: Natriuretic Peptide System as Therapy in Human Preclinical Left Ventricle Dysfunction
Acronym: PPG1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Horng Chen (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Horng Chen, MD, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 05-004027; P01HL076611 (NIH); R01HL084155 (NIH); UL1RR024150 (NIH); NCT00818974 (obsolete NCT alias)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2012-05-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-04

CONDITIONS: Congestive Heart Failure
Keywords: heart failure; diastolic dysfunction; systolic dysfunction; preclinical; natriuretic peptide; B-type natriuretic peptide; cyclic guanosine monophosphate
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo First, then Nesiritide (Arm A) (Experimental): In the first intervention period the subjects received subcutaneous placebo given in the abdomen. After a lead in period of 15 minutes, the acute saline load was administered. There was a 2 week washout period. In the second intervention period, the subjects received subcutaneous nesiritide given in the abdomen. After a lead in period of 15 minutes, the acute saline load was administered.
  Interventions: Drug: Nesiritide; Drug: Placebo; Drug: Saline
- Nesiritide First, then Placebo (Arm B) (Experimental): In the first intervention period the subjects received subcutaneous nesiritide given in the abdomen. After a lead in period of 15 minutes, the acute saline load was administered. There was a 2 week washout period. In the second intervention period, the subjects received subcutaneous placebo given in the abdomen. After a lead in period of 15 minutes, the acute saline load was administered.
  Interventions: Drug: Nesiritide; Drug: Placebo; Drug: Saline

INTERVENTIONS:
Drug: Nesiritide — The first 10 subjects in each group will receive a dose of 5 ug/kg and the next ten subjects will receive 10 ug/kg.
  Other Names: natrecor; human B-type natriuretic peptide (BNP)
Drug: Placebo — The pharmacy created a placebo subcutaneous injection volume to match the volume of the nesiritide dose.
Drug: Saline — Normal saline 0.9% 0.25 ml/kg/min for 60 minutes

SUMMARY:
In congestive heart failure, cardiac output is low, blood pressure is high, and the body becomes congested with fluid. In normal people, when there is high blood pressure, the heart muscle cells secrete a hormone that excretes sodium and water in the urine, reducing blood pressure. The action of this hormone is called the natriuretic response. The purpose of this study is to determine if nesiritide can improve an impaired natriuretic response in subjects with asymptomatic systolic heart failure or asymptomatic diastolic heart failure.

DETAILED DESCRIPTION:
The American Heart Association and the American College of Cardiology define stage B heart failure (HF) as asymptomatic subjects with abnormal heart structure/function. With the advancement of cardiac imaging and biomarkers, abnormal heart structure and function can be detected before the development of symptoms. Stage B HF can represent either diastolic or systolic dysfunction and both are at increased risk of adverse cardiac events and development of symptomatic HF.

The broad objective of this study is to define the integrated cardiorenal response to acute volume expansion (VE) in humans with presystolic dysfunction (PSD), prediastolic dysfunction (PDD), and normal cardiac function. We hypothesized that there is an impaired cardiorenal endocrine response to acute VE in PSD and PDD which is characterized by the lack of appropriate activation of urinary cGMP and urinary sodium excretion. Further, we hypothesized that PSD, PDD, and normal control subjects would respond similarly to exogenous administration B-type natriuretic peptide (BNP).

The natriuretic peptides (NPs) are a family of structurally similar but genetically distinct peptides with vasodilating, natriuretic, renin inhibiting, and lusitropic properties. Acute peptide therapy with brain natriuretic peptide (BNP) infusion has recently been approved by the FDA as a therapeutic strategy for the treatment of acute human decompensated congestive HF. We will determine the effects of acute subcutaneous BNP or placebo administration on the integrated cardiorenal and humoral response to acute sodium load (sodium chloride 0.9% 0.25 ml/kg/min for 1 hour) in three groups of subjects: Group 1 normal controls, Group 2 with PSD, and Group 3 with PDD. Doppler echocardiography and tonometry will be used to measure cardiac and vascular function before and during the sodium load. Renal function studies will assess sodium excretion, renal plasma flow, and glomerular filtration rate at baseline, during, and after the sodium load. Blood will be drawn for humoral analysis including catecholamines, renin, aldosterone, angiotensin II, atrial natriuretic peptide (ANP), BNP, and cyclic guanosine monophosphate (cGMP) at baseline, during, and after the sodium load.

ELIGIBILITY:
Inclusion criteria for normal control group:

* ejection fraction of greater 50%
* normal Doppler diastolic function with no clinical signs or symptoms
* history of cardiovascular and renal disease
* no prior use of any cardiovascular medications.

Inclusion criteria for pre-systolic dysfunction group:

* ejection fraction of less than 40% with no clinical signs or symptoms of congestive heart failure
* ability to perform a 6-minute walk of > 450 meters
* if subjects are not able to walk 450 meters due to pain in hips and knees and not fatigue or shortness of breath, then they will still qualify for the study
* subjects will all be on stable doses of ACE inhibitor for two weeks prior to the active study date
* previously prescribed cardiovascular medications are allowed, however, all medications must be at stable doses two weeks prior to the study date.

Inclusion criteria for pre-diastolic dysfunction group:

* ejection fraction of greater than 50% with moderate or severe diastolic dysfunction as assessed by Doppler echocardiography
* no signs or symptoms of congestive heart failure
* ability to perform a 6-minute walk of > 450 meters
* if subjects are not able to walk 450 meters due to pain in hips and knees and not fatigue or shortness of breath, then they will still qualify for the study
* previously prescribed cardiovascular medications are allowed, however, all medications must be at stable doses two weeks prior to the study date.

Exclusion criteria for all groups:

* myocardial infarction within 3 months of screening
* unstable angina within 14 days of screening, or any evidence of myocardial ischemia
* significant valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* severe congenital heart diseases
* sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* second or third degree heart block without a permanent cardiac pacemaker
* stroke within 3 months of screening, or other evidence of significantly compromised CNS perfusion
* total bilirubin of > 1.5 mg/dL or other liver enzymes >1.5 times the upper limit of normal
* serum creatinine of > 3.0 mg/dL
* serum sodium of < 125 mEq/dL or > 160 mEq/dL
* serum potassium of < 3.5 mEq/dL or > 5.0 mEq/dL
* serum digoxin level of > 2.0 ng/ml
* systolic pressure of < 85 mmHg
* hemoglobin < 10 gm/dl
* other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data
* received an investigational drug within 1 month prior to dosing
* patients with an allergy to iodine
* in the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-02; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] McKie PM, Schirger JA, Costello-Boerrigter LC, Benike SL, Harstad LK, Bailey KR, Hodge DO, Redfield MM, Simari RD, Burnett JC Jr, Chen HH. Impaired natriuretic and renal endocrine response to acute volume expansion in pre-clinical systolic and diastolic dysfunction. J Am Coll Cardiol. 2011 Nov 8;58(20):2095-103. doi: 10.1016/j.jacc.2011.07.042. PMID 22051332

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place between February 2006 and August 2009. All subjects were consented and were seen at the Mayo Clinic in Rochester, MN.
Pre-assignment Details: 63 participants were enrolled in the study, but 5 participants were excluded because they did not meet inclusion criteria. Participants included normal controls, Preclinical Systolic Dysfunction, and Preclinical Diastolic Dysfunction subjects, who were randomized into Placebo First, then Nesiritide (Arm A) and Nesiritide First, then Placebo (Arm B)
Period: First Intervention
Arm/Group | Placebo First, Then Nesiritide (Arm A) | Nesiritide First, Then Placebo (Arm B)
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Placebo First, Then Nesiritide (Arm A) | Nesiritide First, Then Placebo (Arm B)
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Nesiritide (Arm A) | Nesiritide First, Then Placebo (Arm B)
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group (Normals): Healthy volunteers without heart disease
- Preclinical Systolic Dysfunction Group (PSD): Participants with ejection fraction <40% and no heart failure symptoms
- Preclinical Diastolic Dysfunction Group (PDD): Participants with an ejection fraction of > 50% and no heart failure symptoms
- Total: Total of all reporting groups
Arm/Group | Control Group (Normals) | Preclinical Systolic Dysfunction Group (PSD) | Preclinical Diastolic Dysfunction Group (PDD) | Total
Number analyzed (Participants) | 20 | 20 | 18 | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (11) | 65 (12) | 72 (7) | 57.5 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 2 | 9 | 28
  Male | 3 | 18 | 9 | 30
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 18 | 58
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.9 (0.1) | 1.1 (0.2) | 1.1 (0.3) | 1.0 (0.2)
Blood Urea Nitrogen [Mean (Standard Deviation); unit: mg/dL] | 11 (5) | 21 (10) | 23 (6) | 18.2 (8.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
  BMI Categories:
  Underweight = <18.5 Normal weight = 18.5-24.9 Overweight = 25-29.9 Obesity = BMI of 30 or greater
  kg/m^2 | 25 (4) | 31 (5) | 30 (5) | 28.5 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Natriuresis (Urinary Sodium Excretion) in Control Subjects at 60 Minutes After Volume Expansion Compared to Baseline in Response to Placebo Treatment
Description: Value at 60 minutes minus value at baseline.
Time Frame: baseline and 60 minutes
Population: per protocol
Measure: Mean (Standard Error); unit: mEq/min
Groups:
- Control Group: Healthy volunteers without heart disease. Prior to initiation of study, subjects drank water and emptied their bladders to reach an equilibrium, then baseline urine samples were collected. After these samples were collected, all subjects were randomized into Placebo First, then Nesiritide (Arm A) or Nesiritide First, then Placebo (Arm B).
Arm/Group | Control Group
Number analyzed (Participants) | 20
mEq/min | 87.19 (22.26)
Statistical Analysis 1: Comparison: Control Group; Test type: Superiority or Other; p < 0.05, t-test, 1 sided; With Bonferroni correction for multiple comparisons

2. Secondary Outcome: Change in Urinary Cyclic Guanosine Monophosphate (cGMP) in Control Subjects at 60 Minutes After Volume Expansion Compared to Baseline in Response to Placebo Treatment
Description: Value at 60 minutes minus value at baseline
Time Frame: baseline and 60 minutes
Population: intention to treat (ITT)
Measure: Mean (Standard Error); unit: pmol/min
Groups:
- Control Group: Healthy volunteers without heart disease. Prior to initiation of study, subjects drank water and emptied their bladders to reach an equilibrium, then baseline urine samples were collected. After these samples were collected, all subjects were randomized into Placebo First, then Nesiritide (Arm A) and Nesiritide First, then Placebo (Arm B).
Arm/Group | Control Group
Number analyzed (Participants) | 20
pmol/min | 98.23 (34.12)
Statistical Analysis 1: Comparison: Control Group; Test type: Superiority or Other; p < 0.05, rank-sum test; Rank-sum test was used due to non-normality of data with Bonferroni correction for multiple comparisons

3. Secondary Outcome: Change in Natriuresis (Urinary Sodium Excretion) at 30 Minutes in Response to Nesiritide Treatment Compared to Placebo Treatment
Description: Value of natriuresis at 30 min on nesiritide treatment minus value of natriuresis at 30 min on placebo treatment (per subject group). The baseline was not involved in this calculation.
Time Frame: 30 minutes
Population: intention to treat (ITT)
Measure: Mean (Standard Error); unit: mEq/min
Groups:
- Control: Healthy volunteers without heart disease. Prior to initiation of study, subjects drank water and emptied their bladders to reach an equilibrium, then baseline urine samples were collected. After these samples were collected, all subjects were randomized into Placebo First, then Nesiritide (Arm A) or Nesiritide First, then Placebo (Arm B).
- PSD-Preclinical Systolic Dysfunction: Participants with ejection fraction <40% and no heart failure symptoms. Prior to initiation of study, subjects drank water and emptied their bladders to reach an equilibrium, then baseline urine samples were collected. After these samples were collected, all subjects were randomized into Placebo First, then Nesiritide (Arm A) or Nesiritide First, then Placebo (Arm B).
- PDD-Preclinical Diastolic Dysfunction: Participants with an ejection fraction of > 50% and no heart failure symptoms. Prior to initiation of study, subjects drank water and emptied their bladders to reach an equilibrium, then baseline urine samples were collected. After these samples were collected, all subjects were randomized into Placebo First, then Nesiritide (Arm A) or Nesiritide First, then Placebo (Arm B).
Arm/Group | Control | PSD-Preclinical Systolic Dysfunction | PDD-Preclinical Diastolic Dysfunction
Number analyzed (Participants) | 20 | 20 | 18
mEq/min | 440.93 (76.67) | 261.07 (101.60) | 242.82 (68.58)

4. Secondary Outcome: Change in Natriuresis (Urinary Sodium Excretion) at 60 Minutes in Response to Nesiritide Treatment Compared to Placebo Treatment
Description: Value of natriuresis at 60 min on nesiritide treatment minus value of natriuresis at 60 min on placebo treatment (per subject group). The baseline was not involved in this calculation.
Time Frame: 60 minutes
Population: intention to treat (ITT)
Measure: Mean (Standard Error); unit: mEq/min
Arm/Group | Control | PSD-Preclinical Systolic Dysfunction | PDD-Preclinical Diastolic Dysfunction
Number analyzed (Participants) | 20 | 20 | 18
mEq/min | 183.83 (60.60) | 226.89 (101.72) | 41.55 (46.07)

5. Secondary Outcome: Change in Urinary Cyclic Guanosine Monophosphate (cGMP) at 30 Minutes in Response to Nesiritide Treatment Compared to Placebo Treatment
Description: Value of cGMP at 30 min on nesiritide treatment minus value of cGMP at 30 min on placebo treatment (per subject group). The baseline was not involved in this calculation.
Time Frame: 30 minutes
Population: intention to treat (ITT)
Measure: Mean (Standard Error); unit: pmol/min
Arm/Group | Control | PSD-Preclinical Systolic Dysfunction | PDD-Preclinical Diastolic Dysfunction
Number analyzed (Participants) | 20 | 20 | 18
pmol/min | 244.69 (59.09) | 255.31 (59.60) | 353.37 (155.65)

6. Secondary Outcome: Change in Urinary Cyclic Guanosine Monophosphate (cGMP) at 60 Minutes in Response to Nesiritide Treatment Compared to Placebo Treatment
Description: Value of cGMP at 60 min on nesiritide treatment minus value of cGMP at 60 min on placebo treatment (per subject group). The baseline was not involved in this calculation.
Time Frame: 60 minutes
Measure: Mean (Standard Error); unit: pmol/min
Arm/Group | Control | PSD-Preclinical Systolic Dysfunction | PDD-Preclinical Diastolic Dysfunction
Number analyzed (Participants) | 20 | 20 | 18
pmol/min | 303.32 (71.21) | 384.62 (120.47) | 335.29 (90.48)

7. Primary Outcome: Placebo Pre-Treatment Urinary Sodium Excretion After Volume Expansion (UnaV)
Description: Subjects received subcutaneous placebo in the abdomen. After 15 minutes, the acute saline load (volume expansion, VE) was administered. Subjects were asked to empty bladder spontaneously every 30 min (if unable to void every 30 min, a urinary catheter was placed). Adequate bladder emptying was insured by ultrasonography. UNaV was collected at baseline (immediately before VE) and at 30 and 60 min after initiation of VE.
Time Frame: Baseline, 30 min, 60 min
Measure: Mean (Standard Deviation); unit: uEq/min
Arm/Group | Control Group (Normals) | Preclinical Systolic Dysfunction Group (PSD) | Preclinical Diastolic Dysfunction Group (PDD)
Number analyzed (Participants) | 20 | 20 | 18
uEq/min
  Urinary Sodium Excretion (Baseline/Pre-treatment) | 186.6 (67.3) | 255.4 (189.2) | 202.1 (137.5)
  Urinary Sodium Excretion at 30 min | 197.4 (80.8) | 221.0 (118.6) | 187.9 (110.3)
  Urinary Sodium Excretion at 60 min | 211.8 (89.5) | 231.1 (130.8) | 205.0 (130.5)

8. Primary Outcome: Placebo Pre-Treatment Urinary cGMP Excretion After Volume Expansion (UcGMPV)
Description: Subjects received subcutaneous placebo in the abdomen. After 15 minutes, the acute saline load (volume expansion, VE) was administered. Subjects were asked to empty bladder spontaneously every 30 min (if unable to void every 30 min, a urinary catheter was placed). Adequate bladder emptying was insured by ultrasonography. UcGMPV was collected at baseline (immediately before VE) and at 30 and 60 min after initiation of VE.
Time Frame: Baseline, 30 min, 60 min
Measure: Mean (Standard Deviation); unit: pmol/min
Arm/Group | Control Group (Normals) | Preclinical Systolic Dysfunction Group (PSD) | Preclinical Diastolic Dysfunction Group (PDD)
Number analyzed (Participants) | 20 | 20 | 18
pmol/min
  Urinary cGMP Excretion (Baseline/Pre-treatment) | 97.8 (124.8) | 219.5 (188.1) | 245.8 (198.7)
  Urinary cGMP Excretion at 30 min | 154.9 (141.7) | 133.3 (109.9) | 134.4 (114.4)
  Urinary cGMP Excretion at 60 min | 196.0 (182.6) | 134.1 (97.7) | 139.7 (118.6)

9. Primary Outcome: Nesiritide Pre-Treatment Urinary Sodium Excretion After Volume Expansion (UNaV)
Description: Subjects received subcutaneous Nesiritide in the abdomen. After 15 minutes, the acute saline load (volume expansion, VE) was administered. Subjects were asked to empty bladder spontaneously every 30 min (if unable to void every 30 min, a urinary catheter was placed). Adequate bladder emptying was insured by ultrasonography. UNaV was collected at baseline (immediately before VE) and at 30 and 60 min after initiation of VE.
Time Frame: Baseline, 30 min, 60 min
Measure: Mean (Standard Deviation); unit: uEq/min
Arm/Group | Control Group (Normals) | Preclinical Systolic Dysfunction Group (PSD) | Preclinical Diastolic Dysfunction Group (PDD)
Number analyzed (Participants) | 20 | 20 | 18
uEq/min
  Urinary Sodium Excretion (Baseline/Pre-treatment) | 183.9 (58.1) | 232.6 (166.7) | 219.1 (201.7)
  Urinary Sodium Excretion at 30 min | 393.4 (143.4) | 314.7 (225.3) | 303.2 (185.0)
  Urinary Sodium Excretion at 60 min | 650.1 (337.9) | 469.4 (458.9) | 464.8 (272.7)

10. Primary Outcome: Nesiritide Pre-Treatment Urinary cGMP Excretion After Volume Expansion (UcGMPV)
Description: Subjects received subcutaneous Nesiritide in the abdomen. After 15 minutes, the acute saline load (volume expansion, VE) was administered. Subjects were asked to empty bladder spontaneously every 30 min (if unable to void every 30 min, a urinary catheter was placed). Adequate bladder emptying was insured by ultrasonography. UcGMPV was collected at baseline (immediately before VE) and at 30 and 60 min after initiation of VE.
Time Frame: Baseline, 30 min, 60 min
Measure: Mean (Standard Deviation); unit: pmol/min
Arm/Group | Control Group (Normals) | Preclinical Systolic Dysfunction Group (PSD) | Preclinical Diastolic Dysfunction Group (PDD)
Number analyzed (Participants) | 20 | 20 | 18
pmol/min
  Urinary cGMP Excretion (Baseline/Pretreatment) | 130.8 (145.9) | 192.2 (157.3) | 258.0 (176.2)
  Urinary cGMP Excretion at 30 min | 399.6 (252.6) | 388.6 (276.7) | 487.8 (634.0)
  Urinary cGMP Excretion at 60 min | 508.4 (382.3) | 518.7 (578.3) | 475.0 (347.2)

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events from the time of randomization until the completion of the second visit, approximately two months.
Groups:
- Placebo: The pharmacy created a placebo subcutaneous injection volume to match the volume of the nesiritide dose. As this was a cross over study, all participants received placebo and nesiritide.
- Nesiritide: The first 10 subjects in each group received a dose of 5 ug/kg and the next 10 subjects received a dose of 10 ug/kg. As this was a cross over study, all participants received placebo and nesiritide.
Arm/Group | Placebo | Nesiritide
Serious Adverse Events (participants affected / at risk) | 0/58 | 1/58
Other Adverse Events (participants affected / at risk) | 5/58 | 6/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=58) | Nesiritide (N=58)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=58) | Nesiritide (N=58)
re-stenosis (Cardiac disorders) | 0 (0) | 1 (1)
heart palpatations (Cardiac disorders) | 0 (0) | 1 (1)
afibrillation (Cardiac disorders) | 1 (1) | 0 (0)
atypical chest pain (Cardiac disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
hypotension (Cardiac disorders) | 0 (0) | 2 (2)
urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
esophageal reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
* Different baseline characteristics of the three groups of subjects
* Did not define a mechanism for the impaired renal cGMP activation
* Future studies needed to determine effects of chronic nesiritide therapy in preclinical HF.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No